CLINICAL TRIAL: NCT04058925
Title: Cerebral and Skeletal Muscle Oxygenation During Cardiopulmonary Resuscitation as a Predictor of Return of Spontaneous Circulation
Brief Title: Tissue Oxygenation During Cardiopulmonary Resuscitation as a Predictor of Return of Spontaneous Circulation
Status: Completed | Type: Observational
Sponsor: Miha Košir (Other)
Collaborators: University Medical Centre Ljubljana (Other); Community Health Centre Ljubljana (Other)
Responsible Party: Sponsor-Investigator, Miha Košir, Emergency medicine resident, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Other Study IDs: UMC-NIRS/CPR
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Out-Of-Hospital Cardiac Arrest; Near-infrared spectroscopy
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: NIRS device — Application of NIRS electrode to forehead and thenar eminence.

SUMMARY:
The main objective of the trial is to find out if there is correlation between cerebral and skeletal muscle oxygenation values during cardiopulmonary resuscitation and if these values can predict return of spontaneous circulation. The investigators would like to find out which values, first measures, average, maximal, are better predictor of return of spontaneous circulation. All the patients with nontraumatic cardiac arrest in prehospital environment will be enrolled in the study. The measurements will be taken with NIRS device and special electrodes, which will be placed on patient's forehead and thenar eminence od right hand. No ALS procedure will be modified.

DETAILED DESCRIPTION:
Out of hospital cardiac arrest (OHCA) is major cause of morbidity and mortality around the world. Annually there is around 350.000 deaths in the Europe because of OHCA. Despite a great progress in prehospital and emergency medicine in recent years, there is no major increase in surviving OHCA. There are many factors which influence to the end result of OHCA. Till now we still don't know how to predict the outcome of cardiac arrest in early phase of cardiopulmonary resuscitation (CPR).

Today emergency teams use end-tidal CO2 values (etCO2) as an indirect marker of cardiac output and as an auxiliary indicator of return of spontaneous circulation (ROSC). Higher values are also correlated with greater probability of ROSC.

Studies in recent years showed that there could be another method which could help to predict the result of OHCA. Near-infrared spectroscopy (NIRS) is a noninvasive spectroscopic method, which uses light near to infrared electromagnetic spectrum of light. The device can, based on Beer-Lambert law, calculates tissue oxygenation of underlaid tissue. It is also useful in the states, where there is little or even no blood flow (cardiac arrest). NIRS is currently used in operating rooms and ICU, but there is also option to use it in prehospital environment. During cardiac arrest the blood flow through organs is very low or absent. This causes hypoxic-ischemic brain injury and also injury of other vital organs. Based on previous studies with NIRS, we can measure cerebral oxygenation by placing electrodes on patient's forehead. Patients with higher values had greater probability of ROSC. It is presumed, that NIRS values are indirect indicator of coronary perfusion pressure. It is known that higher coronary perfusion pressure is connected with higher oxygen concentration in the brain during cardiac arrest. NIRS can also predict re-arrest even before losing a pulse.

Till today there are no studies which would look for correlation between cerebral and skeletal oxygenation during cardiac arrest.

The investigator's study is monocentric, prospective, observational, nonrandomized taking place at Emergency department of University Medical Centre Ljubljana (UMC Ljubljana). There is also a Basic emergency first aid infirmary (Unit SNMP) of Community Health Centre Ljubljana, which will with it's prehospital units make the measurements. After an eyewitness of cardiac arrest will call on emergency number 112 a medical dispatcher will activate medical team with emergency doctor and send them to the location. Upon arrival the team will start CPR based on ALS protocol. As soon as possible one of team members will put two NIRS electrodes on the patient - one on the patient's forehead and the other on patient's thenar eminence on the hand. ALS protocol will not be modified in any way. The NIRS device (Nonin SenSmart Model X-100) will be turned on till the end of resuscitation or till arrival to the hospital (UMC Ljubljana).

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic cardiac arrest in prehospital environment
* age 18 years or more

Exclusion Criteria:

* age 18 years or less
* pregnancy
* traumatic cause of cardiac arrest
* hypothermia
* drowning
* E-CPR protocol (candidates for ECMO CPR)
* spontaneous circulation upon arrival of emergency team at the scene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult population of city Ljubljana and surrounding municipality is which the emergency first aid is provided by Basic emergency first aid infirmary of Community Health Centre Ljubljana. The area is 1670 km2 big and there are up to 450.000 people.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Correlation between cerebral oxygenation and skeletal oxygenation values. | 30 minutes
  coefficient
First measures cerebral oxygenation and skeletal oxygenation values as a predictor of ROSC. | 1 minute
  percent
Average values of cerebral oxygenation and skeletal oxygenation values as a predictor of ROSC. | 30 minutes
  percent
Absolute change of cerebral oxygenation and skeletal oxygenation values in ROSC and NON-ROSC patients. | 30 minutes
  percent

CONTACTS AND LOCATIONS:
Overall Officials: Matej Podbregar, MD PhD, Principal Investigator — General hospital Celje, Intensive internal medicine therapy unit
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grasner JT, Bottiger BW, Bossaert L; European Registry of Cardiac Arrest (EuReCa) ONE Steering Committee; EuReCa ONE Study Management Team. EuReCa ONE - ONE month - ONE Europe - ONE goal. Resuscitation. 2014 Oct;85(10):1307-8. doi: 10.1016/j.resuscitation.2014.08.001. Epub 2014 Aug 15. No abstract available. PMID 25132474
- [Background] Sasson C, Rogers MA, Dahl J, Kellermann AL. Predictors of survival from out-of-hospital cardiac arrest: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):63-81. doi: 10.1161/CIRCOUTCOMES.109.889576. Epub 2009 Nov 10. PMID 20123673
- [Background] Sandroni C, Cariou A, Cavallaro F, Cronberg T, Friberg H, Hoedemaekers C, Horn J, Nolan JP, Rossetti AO, Soar J. Prognostication in comatose survivors of cardiac arrest: an advisory statement from the European Resuscitation Council and the European Society of Intensive Care Medicine. Resuscitation. 2014 Dec;85(12):1779-89. doi: 10.1016/j.resuscitation.2014.08.011. PMID 25438253
- [Background] Genbrugge C, Meex I, Boer W, Jans F, Heylen R, Ferdinande B, Dens J, De Deyne C. Increase in cerebral oxygenation during advanced life support in out-of-hospital patients is associated with return of spontaneous circulation. Crit Care. 2015 Mar 24;19(1):112. doi: 10.1186/s13054-015-0837-5. PMID 25887259
- [Background] Frisch A, Suffoletto BP, Frank R, Martin-Gill C, Menegazzi JJ. Potential utility of near-infrared spectroscopy in out-of-hospital cardiac arrest: an illustrative case series. Prehosp Emerg Care. 2012 Oct-Dec;16(4):564-70. doi: 10.3109/10903127.2012.702191. Epub 2012 Jul 23. PMID 22823984
- [Background] Cournoyer A, Iseppon M, Chauny JM, Denault A, Cossette S, Notebaert E. Near-infrared Spectroscopy Monitoring During Cardiac Arrest: A Systematic Review and Meta-analysis. Acad Emerg Med. 2016 Aug;23(8):851-62. doi: 10.1111/acem.12980. PMID 27028004
- [Background] Prosen G, Strnad M, Doniger SJ, Markota A, Stozer A, Borovnik-Lesjak V, Mekis D. Cerebral tissue oximetry levels during prehospital management of cardiac arrest - A prospective observational study. Resuscitation. 2018 Aug;129:141-145. doi: 10.1016/j.resuscitation.2018.05.014. Epub 2018 May 12. PMID 29763712
- [Background] Jones S, Chiesa ST, Chaturvedi N, Hughes AD. Recent developments in near-infrared spectroscopy (NIRS) for the assessment of local skeletal muscle microvascular function and capacity to utilise oxygen. Artery Res. 2016 Dec;16:25-33. doi: 10.1016/j.artres.2016.09.001. PMID 27942271
- [Background] Mozina H, Podbregar M. Near-infrared spectroscopy during stagnant ischemia estimates central venous oxygen saturation and mixed venous oxygen saturation discrepancy in patients with severe left heart failure and additional sepsis/septic shock. Crit Care. 2010;14(2):R42. doi: 10.1186/cc8929. Epub 2010 Mar 23. PMID 20331856
- [Background] Schnaubelt S, Sulzgruber P, Menger J, Skhirtladze-Dworschak K, Sterz F, Dworschak M. Regional cerebral oxygen saturation during cardiopulmonary resuscitation as a predictor of return of spontaneous circulation and favourable neurological outcome - A review of the current literature. Resuscitation. 2018 Apr;125:39-47. doi: 10.1016/j.resuscitation.2018.01.028. Epub 2018 Feb 2. PMID 29410191
- [Background] Wik L. Near-infrared spectroscopy during cardiopulmonary resuscitation and after restoration of spontaneous circulation: a valid technology? Curr Opin Crit Care. 2016 Jun;22(3):191-8. doi: 10.1097/MCC.0000000000000301. PMID 27054625
- [Background] Singer AJ, Ahn A, Inigo-Santiago LA, Thode HC Jr, Henry MC, Parnia S. Cerebral oximetry levels during CPR are associated with return of spontaneous circulation following cardiac arrest: an observational study. Emerg Med J. 2015 May;32(5):353-6. doi: 10.1136/emermed-2013-203467. Epub 2014 Mar 24. PMID 24662518
- [Background] Kalkan A, Bilir O, Ersunan G, Ozel D, Tas M, Memetoglu ME. Abdominal oxygen saturation for monitoring return of spontaneous circulation in out-of-hospital cardiac arrest using near infrared spectrophometry. Am J Emerg Med. 2015 Mar;33(3):344-8. doi: 10.1016/j.ajem.2014.11.029. Epub 2014 Nov 28. PMID 25559313
- [Background] Mozina H, Podbegar M. Near-infrared spectroscopy for evaluation of global and skeletal muscle tissue oxygenation. World J Cardiol. 2011 Dec 26;3(12):377-82. doi: 10.4330/wjc.v3.i12.377. PMID 22216373
- [Background] Friess SH, Sutton RM, French B, Bhalala U, Maltese MR, Naim MY, Bratinov G, Arciniegas Rodriguez S, Weiland TR, Garuccio M, Nadkarni VM, Becker LB, Berg RA. Hemodynamic directed CPR improves cerebral perfusion pressure and brain tissue oxygenation. Resuscitation. 2014 Sep;85(9):1298-303. doi: 10.1016/j.resuscitation.2014.05.040. Epub 2014 Jun 16. PMID 24945902
- [Background] Levine RL, Wayne MA, Miller CC. End-tidal carbon dioxide and outcome of out-of-hospital cardiac arrest. N Engl J Med. 1997 Jul 31;337(5):301-6. doi: 10.1056/NEJM199707313370503. PMID 9233867
- [Background] Genbrugge C, De Deyne C, Eertmans W, Anseeuw K, Voet D, Mertens I, Sabbe M, Stroobants J, Bruckers L, Mesotten D, Jans F, Boer W, Dens J. Cerebral saturation in cardiac arrest patients measured with near-infrared technology during pre-hospital advanced life support. Results from Copernicus I cohort study. Resuscitation. 2018 Aug;129:107-113. doi: 10.1016/j.resuscitation.2018.03.031. Epub 2018 Mar 23. PMID 29580958
- [Derived] Kosir M, Mozina H, Podbregar M. Skeletal muscle oxygenation during cardiopulmonary resuscitation as a predictor of return of spontaneous circulation: a pilot study. Eur J Med Res. 2023 Oct 11;28(1):418. doi: 10.1186/s40001-023-01393-z. PMID 37821950